CLINICAL TRIAL: NCT00158951
Title: Device Evaluation of CONTAK(R) RENEWAL 2/4/4HE and EASYTRAK(R) 2: Assessment of Safety and Effectiveness in Heart Failure (DECREASE-HF)
Brief Title: Device Evaluation of Contak Renewal 2and Easytrak 2 - DECREASE-HF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Clinicals0005
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Congestive Heart Failure
Keywords: Left Ventricular Lead; Cardiac Resynchronization Therapy; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: CONTAK RENEWAL 2/4/4HE CRT-D
Device: EASYTRAK 2 Lead

SUMMARY:
The purpose of this clinical investigation is to demonstrate the safety and effectiveness of the CONTAK® RENEWAL™ 2/4/4HE cardiac resynchronization therapy defibrillator (CRT-D) family and EASYTRAK® 2 lead in delivering LV-CRT or BiV-CRT with an LV Offset for patients with heart failure and an indication for an ICD.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, multi-center, randomized, double-blind study design enrolling 360 patients at 57 centers to demonstrate the safety and effectiveness of the therapy, the CONTAK RENEWAL 2/4/4HE devices and the EASYTRAK 2 lead.

ELIGIBILITY:
Inclusion Criteria:

* Meet the general indications for a CRT-D device
* Moderate or severe heart failure, defined as NYHA Class III-IV despite optimal pharmacological heart failure therapy.
* A 12-lead electrocardiogram (ECG) obtained no more than 90 days prior to enrollment documenting a sinus rate > 50 bpm, QRS duration ³ 150 ms, and PR interval £ 320 ms measured from any two leads, and a P-wave duration < 150 ms measured from lead V1
* Creatinine £ 2.5 mg/dL obtained no more than 14 days prior to enrollment
* Left ventricular ejection fraction £ 35% [measured by echo, multiple gated acquisition (MUGA) scan, cardiac catheterization, etc.] no more than 14 days prior to enrollment
* Willing and capable of undergoing a device implant and participating in all testing associated with this clinical investigation
* Have a life expectancy of more than 180 days, per physician discretion
* Age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Right bundle branch block morphology (per World Health Organization Guidelines) on a 12-lead ECG obtained no more than 90 days prior to enrollment.
* Have had previous cardiac resynchronization therapy, a previous coronary venous lead, or meet the general indications for antibradycardia pacing
* Have a neuromuscular, orthopedic, or other non-cardiac condition that prevents normal, unsupported walking
* Have an atrial tachyarrhythmia that is permanent (i.e., does not terminate spontaneously and cannot be terminated with medical intervention) or persistent (i.e., can be terminated with medical intervention, but does not terminate spontaneously) within 180 days prior to enrollment
* Have a hypersensitivity to a 0.7 mg dose of dexamethasone acetate
* Have surgically uncorrected primary valvular heart disease
* Currently requiring dialysis
* Have chronic obstructive pulmonary disease (COPD), defined as FEV1/FVC < 60%
* Have had a myocardial infarct, unstable angina, percutaneous coronary intervention, or coronary artery bypass graft during the 30 days prior to enrollment
* Have hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g., amyloidosis, sarcoidosis)
* Have a mechanical tricuspid prosthesis
* Enrolled in any concurrent study, without Guidant written approval, that may confound the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2003-03; Study Completion 2004-10

PRIMARY OUTCOMES:
Therapy Efficacy: Change in cardiac function at six-months
Therapy Safety: CRT does not increase HF related adverse events at six-months
Device Efficacy; Therapy does not affect ability to detect VF, Stable chronic LV thresholds, R-wave amplitudes and impedances
Device Safety: System complication free rate at six-months, Lead related complication free rate at six-months

SECONDARY OUTCOMES:
Therapy Efficacy: Change in cardiac function and reduced HF symptoms
Therapy Safety: Continuous appropriate pacing
Device Efficacy: Stable chronic LV thresholds, R-wave amplitudes and impedances from those not selected in final programming at six-months

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations in the US, Saint Paul, Minnesota, United States